CLINICAL TRIAL: NCT00712803
Title: A Phase I Dose Comparison Study of the Safety and Immunogenicity of rDEN3-3'Ddelta30, a Live Attenuated Virus Vaccine Candidate for the Prevention of Dengue Serotype 3
Brief Title: Safety of and Immune Response to a Dengue Virus Vaccine (rDEN3-3'Ddelta30) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CIR 252
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): One subcutaneous vaccination (10^3 dose of vaccine) of rDEN3-3'D4delta30 vaccine into the deltoid region of either arm.
  Interventions: Biological: rDEN3-3'D4delta30
- 2 (Experimental): One subcutaneous vaccination (10^5 dose of vaccine or placebo) of rDEN3-3'D4delta30 vaccine into the deltoid region of either arm OR one subcutaneous vaccination (10^1 dose of vaccine or placebo) of rDEN3-3'D4delta30 vaccine into the deltoid region of either arm.
  Interventions: Biological: rDEN3-3'D4delta30

INTERVENTIONS:
Biological: rDEN3-3'D4delta30 — Live attenuated 10^3 dose of rDEN3-3'D4delta30 vaccine.
  Arms: 1
Biological: rDEN3-3'D4delta30 — Live attenuated 10^5 dose of rDEN3-3'D4delta30 vaccine.
  Arms: 2
Biological: rDEN3-3'D4delta30 — Live attenuated 10^1 dose of rDEN3-3'D4delta30 vaccine.
  Arms: 2

SUMMARY:
Dengue fever, which is caused by dengue viruses, is a major health problem in tropical and subtropical regions of the world. The purpose of this study is to evaluate the safety of and immune response to a new dengue virus vaccine in healthy adults.

DETAILED DESCRIPTION:
Dengue viruses cause dengue fever and the more severe dengue hemorrhagic fever/shock syndrome. More than 2 billion people living in tropical and subtropical regions of the world are at risk of dengue virus infection, which is the leading cause of hospitalization and death in children in several tropical Asian countries. This study will evaluate the safety and immunogenicity of a live attenuated dengue virus vaccine called rDEN3-3'D4delta30. This vaccine is derived from rDEN4delta30, another dengue virus vaccine candidate that has been shown to be safe and immunogenic in Phase I and II trials in healthy adults.

There will be two groups in this study. Participants in Group 1 will be randomly assigned to receive rDEN3-3'D4delta30 vaccine or placebo at study entry. The dosing for Group 2 will be determined by a safety review of all participants in Group 1. If less than 90 % of the Group 1 participants seroconvert to DEN3 participants in Group 2 will receive a higher dose of rDEN3-3'D4delta30. If at least 90 % of Group 1 participants seroconvert to DEN3, participants in Group 2 will receive a lower dose of rDEN3-3'D4delta30.

All participants will be required to monitor their temperature three times each day for the first 16 days following each vaccination. Study visits will occur 30 minutes following each vaccination and every other day after vaccination until Day 16, followed by four additional visits at selected days through Day 180. Blood collection, vital signs measurement, and a targeted physical exam will occur at each study visit. Some participants will be asked to undergo a skin biopsy or additional blood collection at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* General good health
* Available for the duration of the study
* Willing to use accepted forms of contraception

Exclusion Criteria:

* Clinically significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease by history, physical examination, or laboratory studies including urinalysis
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, may interfere with the study
* Certain abnormal laboratory values. More information on this criterion can be found in the protocol.
* Medical, work, or family problems as a result of alcohol or illegal drug use within 12 months of study entry
* History of severe allergy or anaphylaxis
* Severe asthma requiring an emergency room visit or hospitalization within 6 months of study entry
* HIV infected
* Hepatitis C virus infected
* Hepatitis B surface antibody positive
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs 30 days prior to study entry. Participants who have used topical or nasal corticosteroids are not excluded.
* Receipt of live vaccine within 4 weeks of study entry
* Receipt of killed vaccine within 2 weeks of study entry
* Absence of spleen
* Plan to travel to an area where dengue virus is common
* Any investigational product within 30 days of study entry
* Other condition that, in the opinion of the investigator, would interfere with the study
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety and immunogenicity, as assessed by neutralizing antibody titers | At 4 weeks and 6 weeks after vaccination
Frequency of vaccine related adverse events as graded by severity | Throughout study

SECONDARY OUTCOMES:
Frequency, quantity, and duration of viremia after a single dose of vaccine | Throughout study
Number of vaccines infected with rDEN3-3'D4delta30 | Throughout study
Infectivity rates, safety, and immunogenicity of a single dose of rDEN3-3'D4delta30 vaccine | Throughout study
Durability of antibody response | At 26 Weeks after vaccination
Obtain an estimate for the Human Infectious Dose-50% (HID50) idf dose dependent infectivity is observed | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research, Johns Hopkins School of Public Health, Washington D.C., District of Columbia
  - Center for Immunization Research, Johns Hopkins University of Public Health, Baltimore, Maryland

REFERENCES:
- [Background] Blaney JE Jr, Hanson CT, Firestone CY, Hanley KA, Murphy BR, Whitehead SS. Genetically modified, live attenuated dengue virus type 3 vaccine candidates. Am J Trop Med Hyg. 2004 Dec;71(6):811-21. PMID 15642976
- [Background] Chaturvedi UC, Shrivastava R, Nagar R. Dengue vaccines: problems and prospects. Indian J Med Res. 2005 May;121(5):639-52. PMID 15937367
- [Background] Guzman MG, Mune M, Kouri G. Dengue vaccine: priorities and progress. Expert Rev Anti Infect Ther. 2004 Dec;2(6):895-911. doi: 10.1586/14789072.2.6.895. PMID 15566333